CLINICAL TRIAL: NCT05904197
Title: Effectiveness of Educational Innovative Gamified Cards About Nephrotic Syndrome for School Age Children on Their Outcomes and Caregivers' Practices
Brief Title: Effectiveness of Educational Gamified Cards About Nephrotic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sara Mustafa Hamza Taha, Assistant Lecturer, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Gamified Health Education
Record Dates: First submitted 2023-05-27; First posted 2023-06-15 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Intervention Model Description: A quasi-experimental (one-group pretest-posttest)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- School age children with nephrotic syndrome and their Caregivers (Other): Children with NS will be expected to have higher knowledge scores about nephrotic syndrome post-intervention than pre-intervention.
  Children with NS will be expected to have higher scores in healthcare-related practices including higher medication adherence post-intervention than pre-intervention.
  Children with NS will be expected to have lower psychosocial problems post-intervention than pre-intervention.
  Caregivers of children with NS will be expected to have higher knowledge scores about nephrotic syndrome post-intervention than pre-intervention.
  Caregivers of children with NS will be expected to have higher scores in health care-related practices post-intervention than pre-intervention.
  Interventions: Other: Gamified Cards about Nephrotic Syndrome

INTERVENTIONS:
Other: Gamified Cards about Nephrotic Syndrome — * The study intervention "Spin to Win - Nephro Cards" will include the following items with simple Arabic language and graphic designation appropriate to children's developmental levels including; nephrotic syndrome, hygiene practices, weight control, fluids, blood pressure control, diet, medication…etc.
  * A spin wheel with numbers and images similar to the educational gamified cards will be designed. Children will request to spin the wheel. After the spin, the educational gamified "Nephro Cards" will reveal and discuss with the child.
  Other Names: Spin to Win - Nephro Cards

SUMMARY:
This study aims to evaluate the effectiveness of educational innovative gamified cards about nephrotic syndrome for school age children on their outcomes and caregivers' practices

DETAILED DESCRIPTION:
Nephrotic Syndrome (NS) is the most common glomerular disorder in children, globally. Eighty percent of NS cases occur in preschool-aged children (less than 6 years of age). The ratio between boys and girls is approximately 2 to 1. It requires long-term treatment and can be recurrent. Steroid responsiveness is one of the critical determinants of the disease course. It has been reported to be 5% for steroid-sensitive NS and 40%-50% for steroid-resistant NS. Although up to approximately 85% of pediatric NS, patients are reportedly sensitive to steroids, most cases relapse, with around half having frequent relapses or becoming steroid-dependent. NS not only compromises the physical health of patients but also affects their psychological health, daily functioning, general well-being, and social functioning. Children with NS are not happy and not satisfied with their lives when compared with their healthy peers. Furthermore, corticosteroid (CS) therapy can cause behavioral abnormalities in children with NS. There was a strong positive correlation between using CS therapy for a long period and the development of psychiatric disorders such as aggression, anxiety, and depression.

Children with NS have unique nutrition support needs. Children should follow a healthy, age-appropriate diet to meet energy requirements and the daily recommended intake of protein. It is recommended to continue to limit sodium, saturated, and trans-saturated fat; as these have been linked to inflammation. Standardized diet recommendations are needed for the regulation of daily energy, sodium, calcium, and vitamin D intakes. Also, the management of the associated conditions and side effects of corticosteroid treatment should be considered. Studies on self-care in childhood NS are very few especially in developing countries (Eid et al, 2020; Rousselet al., 2019). Child education and self-care empowerment are key, which involve both the ability to care for oneself and the activities necessary to achieve, maintain, or promote one's optimal health. Through self-care, various outcomes may be achieved; for example, improved symptom control, coping with the illness, and quality of life (QoL).

In recent years, there has been a lot of attention given to the trend of including game elements in non-gaming facilities. The usage of gamification in education is a massive benefit for motivation, user interaction, and social effects. Gamification is recognized and implemented in diverse areas such as marketing, politics, industry, information technology, fitness exercise, and health . Health researchers and providers have started using gamification apps to deliver medical education online and through mobile apps. Many studies defined the technical term "gamification", it is a mechanism by which game design components are implemented in non-game environments. There are different studies on educational programs that prove the effectiveness of using technologies and gamification with children to promote healthy habits in the short term. Using game-based education, children experience opportunities to solve problems through analytical thinking and improve specific skills through training and adequate feedback. Engagement is also essential for programs designed to promote healthy behaviors.

The nursing role of a child with NS includes relief from edema, enhanced nutritional status, conservation energy, supplying sufficient information about the disease, considering the importance of compliance with the medication and nutritional therapy, and prevention of infection as well as relapse. The nursing Insufficient knowledge, poor compliance to medications, and health-related advice have diverse effects on children with NS including frequent relapse, drug toxicity, higher rates of complications, increased healthcare cost of NS, and high morbidity and mortality rates. In this study, we use empowering school-age children's and their caregivers' education through gamification to support children's self-care.

ELIGIBILITY:
Inclusion Criteria:

* Children with confirmed diagnosis of NS.
* School age child aged between 7 to 12 years old of both gender

Exclusion Criteria:

* Children with associated congenital anomalies.
* Children with mental retardation.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Children's knowledge related to nephrotic syndrome interview questionnaire sheet pre/posttest/ follow-up | through study completion, an average of 6 months.
  This tool will be developed by the researcher in the Arabic language after reviewing the recent related literature to assess the nephrotic children's knowledge related to nephrotic syndrome including the definition of disease, causes, signs and symptoms, nephrotic syndrome specific diet, early signs of infection, oral medication and side effect…etc.
Children's self-reported health-related practices interview questionnaire sheet pre/posttest/ follow-up | through study completion, an average of 6 months.
  This tool will be developed by the researcher in the Arabic language after reviewing the recent related literature to assess the nephrotic children's practices and will cover their reported practices regarding management of NS such as general hygiene practices, regular follow-up measures such as (measuring weight, intake and output, measuring temperature, blood pressure and check protein in urine), administration of medication, proper following of nutrition,.. etc.
Caregivers' knowledge related to nephrotic syndrome interview questionnaire sheet pre/posttest/ follow-up | through study completion, an average of 6 months.
  This tool will be developed by the researcher in the Arabic language after reviewing the recent related literature to assess the nephrotic children's caregivers' knowledge related to nephrotic syndrome this part will include questions about the nature of the disease, its causes and clinical features, drug administration and its side effects, diet, prevention of infections, urine examination at home, related activities and follow up.
Caregivers' self-reported health-related practices interview questionnaire sheet pre/posttest/ follow-up | through study completion, an average of 6 months.
  This tool will be developed by the researcher in the Arabic language after reviewing the recent related literature to assess the nephrotic children's caregivers' practices and will cover their reported practices regarding the management of NS and will be consisted of questions to assess reported practices of caregivers regarding home management of children with NS. This section will include questions regarding practices of the caregivers in situations when the child responds to therapy, receive corticosteroids and has edema or respiratory infections, regular follow-up measures such as (measuring weight, intake and output, measuring temperature, blood pressure and check protein in urine), administration of medication, proper following of nutrition instructions,.. etc.
The Pediatric Symptom Checklist-17 (Psc-17) pre / follow up | through study completion, an average of 6 months.
  It is a psychosocial screen checklist designed to facilitate the recognition of cognitive, emotional behavioral problems. 'The PSC-17 consists of 17 items that are rated as "Never", "Sometimes" or "Often". The PSC helps evaluate how the child is functioning at home, at school, with friends and family, and during other activities in terms of mood and behavior. The PSC helps evaluate how the child is functioning at home, at school, with friends and family, and during other activities in terms of mood and behavior.Caregivers will fill out this tool on behalf of their children
Adherence to Refills and Medications Scale (ARMS) pre / follow up | through study completion, an average of 6 months.
  A validated Arabic version of ARMS will be adopted its 12-item self-reported medication adherence scale consists of two subscales (adherence with filling medications and adherence with taking medications). The adherence with filling medications subscale consists of four items, and the remaining eight items comprise the other subscale (adherence with taking medications).

CONTACTS AND LOCATIONS:
Overall Officials: Fawzia Abusaad, Prof, Principal Investigator — Faculty of Nursing, Mansoura University, Egypt Republik
Locations (1):
- Faculty of Nursing, Mansoura University, Egypt Republik, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhimin L. Self-care in Chinese school-age children with nephrotic syndrome. MCN Am J Matern Child Nurs. 2003 Mar-Apr;28(2):81-5. doi: 10.1097/00005721-200303000-00008. PMID 12629312
- [Background] Krishnamurthy K, Selvaraj N, Gupta P, Cyriac B, Dhurairaj P, Abdullah A, Krishnapillai A, Lugova H, Haque M, Xie S, Ang ET. Benefits of gamification in medical education. Clin Anat. 2022 Sep;35(6):795-807. doi: 10.1002/ca.23916. Epub 2022 Jun 8. PMID 35637557